CLINICAL TRIAL: NCT05996991
Title: Understanding the Impact of Positive, Neutral and Negative Expectation Speech Regarding Manual Therapy Intervention in Patients With Chronic Low Back Pain: a Pilot Study
Brief Title: The Impact of Positive, Neutral and Negative Expectation Speech on Manipulative Therapy Effects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Thais Chaves, Adjunct Professor, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 62827822.2.0000.5504
Record Dates: First submitted 2023-08-04; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Chronic Low-back Pain
Keywords: Placebo Effect; Chronic low-back Pain; Spinal Manipulative Therapy; Expectations; contextual effect
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial with three parallel arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- G1 - Positive Expectation Group + Spinal Manipulative Therapy (Experimental): The participants of G1 will watch a short video (no more than 3 minutes) delivering a positive message regarding SMT. Secondly, a physiotherapist will administer one session of SMT and participants will be re-assessed to investigate the immediate effect of the videos on the pain intensity, global perceived effect of improvement, and expectations. Ultimately, patients will be submitted to a semi-structured interview in which their perceptions about the videos will be investigated.
  Interventions: Other: Positive expectation speech regarding spinal manipulative therapy; Procedure: Spinal Manipulative Therapy
- G2 - Neutral Expectation Group + Spinal Manipulative Therapy (Active Comparator): The participants of G1 will watch a short video (no more than 3 minutes) delivering a neutral message regarding SMT. Secondly, a physiotherapist will administer one session of SMT and participants will be re-assessed to investigate the immediate effect of the videos on the pain intensity, global perceived effect of improvement, and expectations. Ultimately, patients will be submitted to a semi-structured interview in which their perceptions about the videos will be investigated.
  Interventions: Other: Neutral expectation speech regarding spinal manipulative therapy; Procedure: Spinal Manipulative Therapy
- G2 - Negative Expectation Group + Spinal Manipulative Therapy (Active Comparator): The participants of G1 will watch a short video (no more than 3 minutes) delivering a negative message regarding SMT. Secondly, a physiotherapist will administer one session of SMT and participants will be re-assessed to investigate the immediate effect of the videos on the pain intensity, global perceived effect of improvement, and expectations. Ultimately, patients will be submitted to a semi-structured interview in which their perceptions about the videos will be investigated.
  Interventions: Other: Negative expectation speech regarding spinal manipulative therapy; Procedure: Spinal Manipulative Therapy

INTERVENTIONS:
Other: Positive expectation speech regarding spinal manipulative therapy — Patients will watch a short video with positive expectations regarding spinal manipulative therapy.
  Arms: G1 - Positive Expectation Group + Spinal Manipulative Therapy
Other: Neutral expectation speech regarding spinal manipulative therapy — Patients will watch a short video with neutral expectations regarding spinal manipulative therapy.
  Arms: G2 - Neutral Expectation Group + Spinal Manipulative Therapy
Other: Negative expectation speech regarding spinal manipulative therapy — Patients will watch a short video with negative expectations regarding spinal manipulative therapy.
  Other Names: Manual Therapy
  Arms: G2 - Negative Expectation Group + Spinal Manipulative Therapy
Procedure: Spinal Manipulative Therapy — One session of Spinal Manipulative Therapy. The researcher will administer a posterior and inferior push on the opposite anterior superior iliac spine (ASIS) while passively rotating the subject on the side to be manipulated. The spinal manipulations will be repeated four times during a 5-minute period, with impulses oscillating between the right and left ASIS. In addition, we will administrate mobilizations (anterior-posterior central mobilization), applied for 1 minute in each lumbar vertebra (from L5 to L1), using grade I joint mobilization (patients positioned in the ventral decubitus position).
  Other Names: Manual Therapy

SUMMARY:
The objective of this study will be to identify the short-term impact of positive, neutral, or negative speech on pain intensity (primary outcome). The secondary outcomes assessed will be the global perceived effect of improvement, patient's expectations regarding spinal manipulative therapy (SMT) intervention, and perception of empathy in the therapeutic encounter in patients with chronic low back pain (CLBP). This study will enroll 60 participants with CLBP aged between 18 and 60 years.

This is an exploratory randomized clinical trial. The three groups will receive a manual therapy session after watching the video proposed for their group.

First participants will be assessed for pain intensity, low back pain disability, psychosocial aspects, and expectations related to treatment. Secondly, a researcher not involved in the recruitment of patients will randomly allocate the participants into three different groups (G1- group submitted to positive expectation, G2- group submitted to neutral expectation, and G3- group submitted to negative expectation). After the allocation, the participants will watch a short video (no more than 3 minutes) delivering positive, negative, or neutral messages regarding SMT. And finally, a physiotherapist will administer one session of SMT and participants will be re-assessed to investigate the immediate effect of the videos on the pain intensity, global perceived effect of improvement, and expectations.

Ultimately, patients will be submitted to a semi-structured interview in which their perceptions about the videos will be investigated.

Outcomes will be assessed just immediately after one SMT session.

DETAILED DESCRIPTION:
Background: The term "contextual effect" has been used to reinforce the view that the placebo effect should be understood as an effect related to the therapeutic context, and not restricted to the use of inert treatments. Thus, the placebo effect is inherent to any therapeutic context and also can be used to enhance the effects of treatment with active components. There is evidence of the effectiveness of manipulative therapy in the treatment of chronic low back pain (CLBP), however, for most physical therapy interventions, its effect is small. Thus, strategies to enhance the effects of this therapy, such as through the use of context factors, may contribute to better therapeutic outcomes. The literature describes that positively induced expectations can trigger a placebo effect. There are previous studies that investigated the effect of different speech on SMT in patients with chronic neck pain, but there is no study in CLBP. In addition, no previous study investigated further the perceptions of patients regarding the content and perceptions of the videos.

The objective of this study will be to identify the short-term impact of positive, neutral, or negative speech on pain intensity (primary outcome). The secondary outcomes assessed will be the global perceived effect of improvement, patient's expectations regarding spinal manipulative therapy (SMT) intervention, and perception of empathy in the therapeutic encounter in patients with chronic low back pain (CLBP)

Methods: it will be a randomized controlled trial with a blinded assessor. It will be investigated the effect of the use of a hidden conditioning procedure and the induction of positive expectations on pain intensity after the administration of a manipulative therapy approach.

This is an exploratory randomized clinical trial. The three groups will receive one session of SMT after watching the video proposed for their group.

First participants will be assessed for pain intensity, low back pain disability, psychosocial aspects, and expectations related to treatment. Secondly, a researcher not involved in the recruitment of patients will randomly allocate the participants into three different groups (G1- group submitted to positive expectation, G2- group submitted to neutral expectation, and G3- group submitted to negative expectation). After the allocation, the participants will watch a short video (no more than 3 minutes) delivering positive, negative, or neutral messages regarding SMT. And finally, a physiotherapist will administer one session of SMT and participants will be re-assessed to investigate the immediate effect of the videos on the pain intensity, global perceived effect of improvement, and expectations. Ultimately, patients will be submitted to a semi-structured interview in which their perceptions about the videos will be investigated. It will help to understand if the content of the videos actually causes an impact on the expectations of the patients.

The main hypothesis of this study is that the group submitted to the positive expectation speech will have a higher hypoalgesic effect, greater perception of improvement, and higher expectations regarding SMT than the other groups immediately post-treatment.

Outcomes will be assessed just immediately after one SMT session.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who report non-specific CLBP (in which the specific nociceptive source cannot be identified, confirmed by a medical assessment) for at least three months duration;
2. Age ranged from 18 years to 60 years
3. Baseline pain intensity score ≥3 on a Numeric Pain Rating Scale (NPRS) (because of the measurement error > 2 reported for the NPRS);
4. Patients able to speak and understand Portuguese well to fill out the questionnaires.

Exclusion Criteria:

1. Previous poor experiences with SMT through the application of a brief screening questionnaire
2. Pregnancy
3. Specific low back pain disorders like radiculopathy or lumbar stenosis or chronic degenerative disorders, i.e., uncontrolled cardiovascular, metabolic, or systemic diseases, neurological or psychiatric diseases, and stroke sequelae
4. Undergoing other therapeutic interventions for chronic pain and low back pain (including surgeries) in the last 3 months
5. Presence of contraindications to SMT

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | one-hour after the baseline assessment
  The Numeric Pain Rating Scale (NPRS) will be used to assess pain intensity in this trial and consists in a sequence of numbers from zero to ten, in which zero represents "no pain" and 10 represents "worst pain imaginable"

SECONDARY OUTCOMES:
Global Perceived Effect (GPE) of Improvement | one-hour after the baseline assessment
  The GPE of improvement used for this trial is an 11-point scale that ranges from "-5" ("vastly worse") through zero ("no change") to "+5" ("completely recovered") and patients are asked: "Compared to when this episode first started, how would you describe your orofacial pain these days?". A higher score indicates higher perception of recovery from the condition.
Low-back Pain (LBP) Expectation Scale | one-hour after the baseline assessment
  The LBP Expectation Scale assesses the patient's previous expectation that the LBP will improve. The participant is asked to respond using an 11-point scale, ranging from zero to ten, where zero represents "no chance" and ten represents "very likely".
Treatment Expectations in Chronic Pain Scale (TEC) | one-hour after the baseline assessment
  The TEC scale is a self-report questionnaire measuring patients' ideal and predicted expectations. The scale has 9 items which were designed to measure two aspects of expectations, namely process and outcome expectations. Instructions are as follows: 'The following questions are about your expectations of the treatment you will receive for your chronic pain. For each question, please check the box that best corresponds to (1) what you ideally hope will happen (in an ideal world, what would you want to happen) during your health care appointment(s) and (2) what you realistically expect will happen (in real life, what do you expect will actually happen) during your health care appointment(s). For each item, patients are asked to select the extent to which they agree with the statement on a 5-point scale (1 = strongly disagree to 5 = strongly agree) in terms of their ideal and predicted expectations. Each item is thus scored twice by participants.
Empathy - Care Scale | one-hour after the baseline assessment
  The Consultation and Relational Empathy (CARE) Measure is a person-centred process measure that was developed and researched at the Departments of General Practice in Glasgow University and Edinburgh University. The CARE Measure is a quick (only 10 questions), clear and easy to complete patient-completed questionnaire. It measures empathy in the context of the therapeutic relationship during a one-on-one consultation between a clinician and a patient. The score of the CARE ranges from 10 to 50. Higher the score, higher the perceived quality of the encounter with healthcare professionals.

CONTACTS AND LOCATIONS:
Overall Officials: Thais C Chaves, PHD, Study Chair — Federal University of São Carlos - UFSCar
Locations (1):
- Federal University of São Carlos - Department of Physical Therapy, São Carlos, São Paulo, Brazil